CLINICAL TRIAL: NCT06944028
Title: Evaluation of Selective and Stepwise Excavation in Young Permanent Teeth With Deep Caries Lesions (SELECT): A Randomized Controlled Trial in a Practice-Based Research Network
Brief Title: Evaluation of Selective and Stepwise Excavation in Young Permanent Teeth With Deep Caries Lesions.
Acronym: SELECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Folktandvården Stockholms län AB (Other Government); Praktikertjanst AB (Other)
Responsible Party: Principal Investigator, Maria Anderson, Dr, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2024-03717-01; selective excavation (Other: Karolinska Institutet); SELECT (Other: Folktandvården Stockholms län AB)
Record Dates: First submitted 2025-02-06; First posted 2025-04-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-04

CONDITIONS: Dental Caries; Dental Cavities
Keywords: SELECT; stepwise excavation; selective excavation; deep dental caries lesions; young permanent teeeth
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Masking Description: The statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selective excavation (Experimental): One visit procedure
  Interventions: Procedure: Selective excavation
- Stepwise excavation-two visit procedure (Active Comparator): Two-visit procedure
  Interventions: Procedure: Stepwise excavation

INTERVENTIONS:
Procedure: Selective excavation — Partial removal of carious dentine, soft carious tissue is intentionally left over the pulp to avoid exposure. The peripheral enamel and dentine are prepared to hard dentine, and a permanent restoration is placed on the tooth.
  Arms: Selective excavation
Procedure: Stepwise excavation — Partial removal of carious dentine is performed, soft dentine is intentionally left over the pulp to avoid exposure. The peripheral enamel and dentine are prepared to hard dentine, application of a provisional restoration. After approximately 3-5 months, the provisional restoration is removed, and any remaining carious dentine is further removed until firm dentine is reached. A permanent restoration is then applied.
  Arms: Stepwise excavation-two visit procedure

SUMMARY:
The purpose of this clinical trial is to evaluate and compare the outcomes of selective carious tissue removal versus stepwise carious tissue removal in young permanent teeth with deep carious lesions. The primary follow-up will be conducted 1 year after treatment to assess success. A secondary follow-up will take place 3 years post-treatment, utilizing data from dental registries and dental records. The study is a randomized controlled trial conducted within a practice-based research network.

DETAILED DESCRIPTION:
The SELECT compares selective carious tissue removal and stepwise excavation in young permanent teeth with deep carious lesions. Unlike the traditional approach of total caries excavation-still widely practiced by dentists-the study implements minimally invasive methods in clinical settings. Conducted within a practice-based research network (PBRN), the study ensures that its findings are highly relevant to real-world clinical environments. Targeting young permanent teeth, a population critical for long-term dental health, the study has a robust randomized controlled trial (RCT) design. Its long follow-up period includes a clinical assessments at 1 year, and at 3 years using dental registry data/dental records. The focus on minimally invasive techniques aligns with contemporary trends in conservative dentistry, and the findings have the potential to inform future guidelines, advancing evidence-based and sustainable treatment practices.

Aim: The aim of the SELECT study is to compare the clinical and long-term outcomes of selective carious tissue removal versus stepwise excavation in managing deep carious lesions in young permanent teeth. The study aims to determine which method is more effective in preserving tooth vitality, reducing complications, and supporting sustainable dental health. The implementation of minimally invasive methods in routine dental practice is a key component of this study, emphasizing the importance of patient-centered and less invasive care.

Selection of participants: Participants will be recruited through the PBRN and all eligible patients will be considered if they comply with the clearly defined inclusion and exclusion criteria.

Statistical plan and data analysis: The sample size calculations is based on the statistical power to reject the null hypothesis H0" No difference between treatment types" at a 5% risk level of type I error. The sample size for each treatment group is determined to be 333 participants based on the primary outcome, with a primary follow-up period of 1 to 1,5 year including an attrition rate of 20%. The success probability for stepwise excavation is set at 90%, with a risk difference of +6 percentage points for selective excavation. The study is powered with a type-I error of 5% and a type-II error of 20%. For the follow-up data after 2-3 years, a base success probability of 80% for stepwise excavation was assumed and a risk difference of +10% for selective excavation rending for a sample size of 392 patients. The outcome will be a vital tooth without pain as a binary variable indicating a successful or unsuccessful treatment and a logistic regression analysis will be performed.

Randomization: Only one deep caries lesion per participant will be randomized. The trial will use block randomization.

Blinding: Blinding of the dental team performing the dental treatment or the patient is not possible as there is a one-visit or a two-visit procedure. The statistical analyses will be performed blinded.

Discontinuation and withdrawal: If a patient does not show up for an examination or treatment an effort will be made to reschedule for the visit and finding the reason for not showing up. But the participation is on a voluntary basis and the participant can chose to leave the study at any time. To facilitate the follow-up examination, there is some flexibility in the follow up period. If the patient fail to attend the scheduled appointment, at least one more appointment will be offered and preceded with a phone-call. Loss of follow up has been accounted for in the calculation of sample size

ELIGIBILITY:
Inclusion Criteria:

Children aged 8- 19 years (last December the year they turn 19 years) A fully erupted molar or pre-molar teeth with dental caries (class I or class II) extending to more than 2/3 of the dentine thickness (and on the bitewing radiograph showing a radiodense zone separating the pulp from the demineralized dentine).

Bitewing radiograph has been taken as part of the ordinary dental examination Available for recall at least for 1 year.

Exclusion Criteria:

Extraction is planned of the tooth with deep caries in the future with expected spontaneous gap closure.

If the carious tooth shows sign or symptoms of irreversible pulp pathology or loss of vitality including:

* Presence of a sinus tract (fistula)
* Tenderness to percussion
* Buccal tenderness
* Severe sensitivity
* Evidence of pathology on a periapical radiograph (if radiograph is clinically justified and performed)
* No written informed consent.
* Medical condition requiring special considerations with regard of the dental management
* Dental treatment cannot be performed adequate due to lack cooperation

Ages: 8 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 666 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Sustained tooth vitality | 1-1,5 years after baseline
  The examining dentist will aggregate a combination of clinical tests and radiographic findings that need to be fulfilled, to assess the outcome: sustained tooth vitality.
  All assessments will be recorded separately. The following measures will be recorded: positive response to cold test, absence of fistula or abscess, absence of tenderness on percussion, no evidence of pulp necrosis based on a periapical radiograph (if clinically justified and performed), no root filling.
  Additionally, the examining dentist will document which tests have been performed to justify the assessment.

SECONDARY OUTCOMES:
Health economic | Up to 3 years (after baseline)
  Costs (direct and indirect)
Quality of life (Qol) | 1 -1,5 years after baseline
  The EQ-5D-Y will be used to assess QoL. The EQ-5D-Y is a generic health-related quality of life (HRQoL) measure developed for youth from 8 years old that comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS) 0-100 where higher score means better outcome. For more information: https://euroqol.org/wp-content/uploads/2023/11/Userguide-EQ5D-Y-23-07.pdf
No pain from tooth | 1-1,5 years after baseline
  Absence of pain from the tooth as reported by the patient and documented by the examining dentist.
Sustained tooth without root canal treatment | Up to 3 years (after baseline)
  Will be determined by the presence by a sustained tooth without root canal treatment at the follow up assessment
Tooth survival | Up to 3 years (after baseline)
  Tooth still present at the follow-up assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Folktandvården Stockholm, Stockholm, Sweden